CLINICAL TRIAL: NCT07204925
Title: Towards Efficient Personalization of Computerized Lower Limb Prostheses Via Reinforcement Learning in a Clinical Setup - Patient Study
Brief Title: Towards Efficient Personalization of Computerized Lower Limb Prostheses Via Reinforcement Learning in a Clinical Setup - Group 1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: North Carolina State University (Other)
Collaborators: Arizona State University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, He Huang, Professor, North Carolina State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 28186; U.S. NIH 1R01HD116422-01A1 (Other Grant/Funding Number: National Institute of Health)
Record Dates: First submitted 2025-09-02; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Transfemoral Amputation
Keywords: Powered prosthesis legs; control parameter personalization; reinforcement learning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: During the evaluation trial, the participants and evaluators are blinded on how the personalized parameters are decided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Tuning expert without RISE (Active Comparator): Tuning experts decide the control parameters based on their knowledge about the powered prosthetic device and patients' feedback
  Interventions: Device: Manual personalization of the prosthetic leg by tuning experts
- Tuning expert with RISE (Active Comparator): The control parameters of the prosthetic legs are decided by tuning experts with the help of the developed RISE system
  Interventions: Device: RISE guided personalization of prosthetic legs by tuning experts
- Prosthetists with RISE (Active Comparator): Control parameters of the prosthetic leg are decided by prosthetists, who are not familiar with the prosthetic leg prototype, with the RISE system.
  Interventions: Device: RISE guided personalization of prosthetic legs by prosthetists

INTERVENTIONS:
Device: RISE guided personalization of prosthetic legs by tuning experts — The personalization procedure is conducted by tuning experts based on the recommendation of RISE system
  Arms: Tuning expert with RISE
Device: RISE guided personalization of prosthetic legs by prosthetists — The control parameters of the prosthetic leg prototype is decided by prosthetists without detailed knowledge about the prosthetic leg with the help of developed RISE system
  Arms: Prosthetists with RISE
Device: Manual personalization of the prosthetic leg by tuning experts — The control parameters of the prosthetic legs are decided by tuning experts based on their knowledge of the prosthetic leg prototypes and patients' response.
  Arms: Tuning expert without RISE

SUMMARY:
The goal of this clinical trial is to understand the feasibility and effectiveness of using reinforcement learning to personalize robotic prosthetic legs (an experimental prototype) for unilateral transfemoral amputees. The main questions it aims to answer are:

* With the developed RL-based Recommendation Interfacing System (RISE), clinicians are able to personalize prosthetic legs faster compared with existing manual personalization procedures.
* With the developed RL-based Recommendation Interfacing System (RISE), clinicians are able to personalize prosthetic legs without detailed knowledge about how the prosthetic legs are controlled.
* Patients perform better when the prosthetic legs are personalized with RISE system compared with the ones personalized manually Researchers will compare two arms (RISE guided personalization and manual personalization) to see if the tuning speed will increase and if patients can perform better.

Participants will go through the standard prosthetic fitting procedures, such as alignment adjustment, then they will experience repeated prosthesis personalization procedures conducted by tuning specialists without RISE, tuning specialists with RISE, and prosthetists (without tuning expertise) with RISE on different types of terrains. In the end, the participants will go through a testing trial, in which they will experience the prototype personalized through the three different approaches without knowing how the control parameters are decided. Their walking performance will be recorded. It is expected that the participants will visit the testing site 8 times, which including alignment (1 visit), three personalization procedures (twice for each), and one testing trial (1-2 visits).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral amputees between 18-75 with K level three or higher
* More than one year after amputation
* Using current prosthetic socket and leg for more than three months
* No major skin issues on the residual limb for more than six months
* Can walk for more than 4 minutes continuously without any other assistive devices

Exclusion Criteria:

* Have very short residual thighs (the length of the residual limb is <15% of the length of the unimpaired limb)
* Are <1.50m in height or >116Kg in weight (who would not fit our prosthesis or the PowerKnee)
* Have cognitive, visual, audio impairments that would affect their ability to give informed consent or to follow simple Instructions during the experiments
* Have any significant co-morbidity that interferes with the study (e.g. stroke, pacemaker placement, pain, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
Total personalization time | During the visit arranged for personalization
  Time needed to finish the personalization of the prosthetic leg

SECONDARY OUTCOMES:
Walking speed | During the last visit for evaluation
  The walking speed of the participants when the prosthetic leg is personalized using one of the three personalization procedures
Step length | During the last visit for evaluation
  Length of step when the participant walking with the prosthetic leg, of which control parameters are decided by one of the three personalization approaches.
foot elevation | during the last visit for evaluation
  Maximum height of the foot during swing when the control parameters of the prosthetic legs are decided by one of the three personalization procedures

CONTACTS AND LOCATIONS:
Overall Officials: He (Helen) Huang, PhD, Principal Investigator — NC State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Based on the requirement of local IRB, we will not share IPD information with other researchers and only deidentified data will be shared.

DOCUMENTS (1):
  • Informed Consent Form (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT07204925/ICF_000.pdf